CLINICAL TRIAL: NCT01526928
Title: A Phase 1/2, Open-Label, Safety, Pharmacokinetic and Preliminary Efficacy Study of Oral Rociletinib in Patients With Previously Treated Mutant EGFR Non-Small Cell Lung Cancer (NSCLC)
Brief Title: Study to Evaluate Safety, Pharmacokinetics, and Efficacy of Rociletinib (CO-1686) in Previously Treated Mutant Epidermal Growth Factor Receptor (EGFR) in Non-Small Cell Lung Cancer (NSCLC) Patients
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Clovis Oncology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CO-1686-008
Record Dates: First submitted 2012-01-31; First posted 2012-02-06 (Estimated); Results first posted 2020-01-06 (Actual); Last update posted 2020-08-04 (Actual); Status verified 2020-07

CONDITIONS: Locally Advanced or Metastatic Non Small Cell Lung Cancer
Keywords: cancer; metastatic; locally advanced; lung; non-small cell lung cancer; NSCLC; epidermal growth factor receptor; EGFR; T790M; CO-1686; unresectable; recurrent; EGFR-directed therapy; irreversible EGFR inhibitor; TIGER; Rociletinib
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Neoplasms; Neoplasm Metastasis; Recurrence | interventions — rociletinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- Rociletinib <900 mg BID FB formulation (Experimental): Rociletinib free base (FB) dose <900 mg twice a day (BID)
  Interventions: Drug: Rociletinib
- Rociletinib 900 mg BID FB formulation (Experimental): Rociletinib free base (FB) dose 900 mg twice a day (BID)
  Interventions: Drug: Rociletinib
- Rociletinib 500 mg BID HBr formulation (Experimental): Rociletinib hydrobromide (HBr) dose 500 mg twice a day (BID)
  Interventions: Drug: Rociletinib
- Rociletinib 625 mg BID HBr formulation (Experimental): Rociletinib hydrobromide (HBr) dose 625 mg twice a day (BID)
  Interventions: Drug: Rociletinib
- Rociletinib 750 mg BID HBr formulation (Experimental): Rociletinib hydrobromide (HBr) dose 750 mg twice a day (BID)
  Interventions: Drug: Rociletinib
- Rociletinib 1000 mg BID HBr formulation (Experimental): Rociletinib hydrobromide (HBr) dose 1000 mg twice a day (BID)
  Interventions: Drug: Rociletinib

INTERVENTIONS:
Drug: Rociletinib — Phase 1: Rociletinib <900 mg BID FB will be administered in escalating dosages in a period of 21-day cycles
  Other Names: CO-1686
  Arms: Rociletinib <900 mg BID FB formulation
Drug: Rociletinib — Phase 1: Rociletinib 900 mg BID FB will be administered in escalating dosages in a period of 21-day cycles
  Other Names: CO-1686
  Arms: Rociletinib 900 mg BID FB formulation
Drug: Rociletinib — Phase 1: Rociletinib 500 mg BID HBr will be administered in escalating dosages in a period of 21-day cycles
  Phase 2: Rociletinib 500 mg BID HBr will be administered daily
  Other Names: CO-1686
  Arms: Rociletinib 500 mg BID HBr formulation
Drug: Rociletinib — Phase 1: Rociletinib 625 mg BID HBr will be administered in escalating dosages in a period of 21-day cycles
  Phase 2: Rociletinib 625 mg BID HBr will be administered daily
  Other Names: CO-1686
  Arms: Rociletinib 625 mg BID HBr formulation
Drug: Rociletinib — Phase 1: Rociletinib 750 mg BID HBr will be administered in escalating dosages in a period of 21-day cycles
  Phase 2: Rociletinib 750 mg BID HBr will be administered daily
  Other Names: CO-1686
  Arms: Rociletinib 750 mg BID HBr formulation
Drug: Rociletinib — Phase 1: Rociletinib 1000 mg BID HBr will be administered in escalating dosages in a period of 21-day cycles
  Phase 2: Rociletinib 1000 mg BID HBr will be administered daily
  Other Names: CO-1686
  Arms: Rociletinib 1000 mg BID HBr formulation

SUMMARY:
Rociletinib is a novel, potent, small molecule irreversible tyrosine kinase inhibitor (TKI) that selectively targets mutant forms of the epidermal growth factor receptor (EGFR) while sparing wild-type (WT) EGFR. The purpose of the study is to evaluate the pharmacokinetic (PK) and safety profile of oral rociletinib; to determine the maximum tolerated dose (MTD) and/or recommended Phase 2 dose (RP2D) of oral rociletinib; to assess the safety and efficacy of rociletinib in previously treated NSCLC patients known to have the T790M EGFR mutation.

DETAILED DESCRIPTION:
Lung cancer remains the most common cancer worldwide with non-small cell lung cancer accounting for 85% of cases. Cytotoxic chemotherapy has been the mainstay of patients with NSCLC; however, survival rates remain low and toxicity is significant. Molecularly targeted therapies have proven to be superior to chemotherapy for NSCLC patients whose tumors have mutations in EGFR. Recent studies have established tyrosine kinase inhibitors (TKIs) as the gold standard for treating EGFR-mutation-positive NCSLC. However, patients on TKIs eventually progress, and in approximately 50% of cases, progression is due to development of an additional mutation called T790M. There are currently no approved therapies for patients who progress on TKIs. Rociletinib may provide an effective therapy for a patient population with few alternative treatment options. Nonclinical data demonstrate that rociletinib inhibits T790M. It is anticipated that rociletinib may promote cell death in tumor cells with the T790M mutation, thus providing possible therapeutic benefit in patients who have developed T790M-mediated resistance to first generation TKIs.

This is a two-part, open-label study of oral rociletinib administered daily in previously treated NSCLC patients who have documented evidence of an activating mutation in the EGFR gene and have failed treatment with an EGFR inhibitor such as erlotinib, gefitinib or afatinib.

This study will include 2 parts:

Phase 1: Dose-escalation Period with 21-day cycles; optional Treatment Extension Period starting on Day 22

Phase 2: Evaluation of activity and safety in patients with the T790M EGFR mutation who have:

Cohort A - Progressed on EGFR directed therapy (irrespective of the number and order of previous lines of NSCLC therapy) or Cohort B - Progression on the first single agent EGFR directed therapy received and also had no more than one previous line of chemotherapy or Cohort C - Patients with discordance between local (T790M positive) and central (T790M negative) T790M results, or had no central test result due to inadequacy of the tissue specimen and known to be T790M positive by local test

ELIGIBILITY:
Inclusion Criteria -

All patients must meet the following inclusion criteria:

1. Metastatic or unresectable locally advanced NSCLC
2. Evidence of a tumor with one or more EGFR mutations excluding exon 20 insertion
3. Biopsy of either primary or metastatic tumor tissue within 60 days of dosing
4. Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1
5. Minimum age of 18 years
6. Adequate hematological and biological function
7. Written consent on an IRB/IEC-approved Informed Consent Form (ICF) prior to any study-specific evaluation

Phase 2 Cohorts must also meet the following inclusion criteria:

* Disease progression confirmed by radiologic assessment while on treatment with EGFR- TKI Or
* Disease progression confirmed by radiologic assessment while on treatment with the first single agent EGFR TKI and
* Documented evidence of T790M mutation in EGFR following disease progression on the first single agent EGFR TKI.
* Measureable disease according to RECIST Version 1.1

Exclusion Criteria -

Any of the following criteria will exclude patients from study participation:

1. Documented evidence of an Exon 20 insertion activating mutation in the EGFR gene
2. Active second malignancy
3. Known pre-existing interstitial lung disease
4. Patients with Leptomeningeal carcinomatosis are excluded. Other CNS metastases are only permitted if treated, asymptomatic and stable (not requiring steroids for at least 4 weeks prior to start of study treatment).
5. Treatment with prohibited medications less than or equal to 14 days prior to treatment with rociletinib
6. Patients who are currently receiving treatment with any medications that have the potential to prolong the QT interval and the treatment cannot be either discontinued or switched to a different medication before starting rociletinib
7. Prior treatment with rociletinib or other drugs that target T790M positive mutant EGFR with sparing of wild type EGFR
8. Certain cardiac abnormalities or history
9. Non-study related surgical procedures less than or equal to 7 days prior to administration of rociletinib
10. Females who are pregnant or breastfeeding
11. Refusal to use adequate contraception for fertile patients (females and males) for 12 weeks after the last dose of rociletinib
12. Presence of any serious or unstable concomitant systemic disorder incompatible with the clinical study
13. Any other reason the investigator considers the patient should not participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 612 (Actual)
Dates: Start 2012-03-27 (Actual); Primary Completion 2018-07-03 (Actual); Study Completion 2018-08-27 (Actual)

CONTACTS AND LOCATIONS:
Locations (49):
- United States (39):
  - City of Hope National Medical Center, Duarte, California
  - Compassionate Care Research Group, Inc., Fountain Valley, California
  - University of Southern California, Norris Comprehensive Cancer Center, Los Angeles, California
  - Samuel Oschin Cancer Center, Los Angeles, California
  - University of California, Irvine, Orange, California
  - University of California Davis Medical Center, Sacramento, California
  - UCLA Health System, Santa Monica, California
  - Stanford Cancer Institute, Stanford, California
  - East Valley Hematology and Oncology Medical Group, Inc., Whittier, California
  - The Oncology Institute of Hope and Innovations, Whittier, California
  - University of Colorado Anschutz Medical Campus, Aurora, Colorado
  - Georgetown University Hospital, Washington D.C., District of Columbia
  - Sylvester Comprehensive Cancer Center/UMHC, Miami, Florida
  - Florida Hospital Cancer Institute, Orlando, Florida
  - University Cancer & Blood Center, Athens, Georgia
  - University of Chicago Medical Center, The Duchossois Center for Advanced Medicine, Chicago, Illinois
  - University of Maryland, Baltimore, Maryland
  - Mass General Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Saint Joseph Mercy Hospital, Ann Arbor, Michigan
  - Karmanos Cancer Care Institute, Detroit, Michigan
  - Regional Cancer Care Associates, Morristown, New Jersey
  - Regional Cancer Center, New Brunswick, New Jersey
  - Roswell Park Cancer Institute, Buffalo, New York
  - Monter Cancer Center, Lake Success, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - University of Cincinnati Medical Center, Cincinnati, Ohio
  - Ohio State University, Comprehensive Cancer Center, Columbus, Ohio
  - Tulsa Cancer Institute, Tulsa, Oklahoma
  - Providence CancerCenter Oncology and Hematology Care Clinic-Eastside Portland, Portland, Oregon
  - Perelman Center for Advanced Medicine, Philadelphia, Pennsylvania
  - University of Pittsburgh Cancer Institute (UPMC), Div. of Medical Oncology, Pittsburgh, Pennsylvania
  - Vanderbilt University, Nashville, Tennessee
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - MD Anderson Cancer Center, Houston, Texas
  - Huntsman Cancer Institute, Salt Lake City, Utah
  - Virginia Cancer Specialists, PC, Fairfax, Virginia
  - Swedish Cancer Institute, Seattle, Washington
  - University of Washington, Seattle, Washington
- Australia (2):
  - Chris O'Brien Lifehouse, Camperdown, New South Wales
  - Peter MacCallum Cancer Centre, East Melbourne
- France (7):
  - Centre Hospitalier Universitaire de Grenoble, Grenoble, Auvergne-Rhône-Alpes
  - Centre Léon Bérard, Lyon, Auvergne-Rhône-Alpes
  - Centre Antoine Lacassagne, Nice, Provence-Alpes-Côte d'Azur Region
  - Centre François Baclesse, Caen
  - Centre Hospitalier Intercommunal Créteil, Créteil
  - Centre Hospitalier Régional Universitaire de Lille, Lille
  - Institut Gustave Roussy, Villejuif
- Med University Gdansk, Gdansk, Poland

REFERENCES:
- [Derived] Krug AK, Enderle D, Karlovich C, Priewasser T, Bentink S, Spiel A, Brinkmann K, Emenegger J, Grimm DG, Castellanos-Rizaldos E, Goldman JW, Sequist LV, Soria JC, Camidge DR, Gadgeel SM, Wakelee HA, Raponi M, Noerholm M, Skog J. Improved EGFR mutation detection using combined exosomal RNA and circulating tumor DNA in NSCLC patient plasma. Ann Oncol. 2018 Mar 1;29(3):700-706. doi: 10.1093/annonc/mdx765. PMID 29216356
- [Derived] Sequist LV, Soria JC, Goldman JW, Wakelee HA, Gadgeel SM, Varga A, Papadimitrakopoulou V, Solomon BJ, Oxnard GR, Dziadziuszko R, Aisner DL, Doebele RC, Galasso C, Garon EB, Heist RS, Logan J, Neal JW, Mendenhall MA, Nichols S, Piotrowska Z, Wozniak AJ, Raponi M, Karlovich CA, Jaw-Tsai S, Isaacson J, Despain D, Matheny SL, Rolfe L, Allen AR, Camidge DR. Rociletinib in EGFR-mutated non-small-cell lung cancer. N Engl J Med. 2015 Apr 30;372(18):1700-9. doi: 10.1056/NEJMoa1413654. PMID 25923550

RESULTS

PARTICIPANT FLOW:
Recruitment Details: There were 612 patients who received rociletinib-111 enrolled in Phase 1 and 501 enrolled in Phase 2. The Phase 1 component of the study was conducted at 8 study sites in the US, Australia, and France. Phase 2 was conducted at 49 study sites in the US, France, Poland, and Australia.
Groups:
- Rociletinib <900 mg BID FB Capsules: Rociletinib free base (FB) dose <900 mg twice a day (BID). FB doses tested ranged from 150 mg once a day (QD) up to 900 mg twice a day (BID). This arm also includes a 400 mg three times a day (TID) dose. Rociletinib FB capsules were administered in Phase 1 only (until November 2013) and were provided in 50 mg or 150 mg white capsules. Patients were instructed to take each dose with 8 oz (240 mL) of water and with a meal or within 30 minutes after a meal. Patients received rociletinib in 21-day treatment cycles and were treated until there was progression by RECIST v1.1, clinical tumor progression, or unacceptable toxicity, or other discontinuation criteria were met. Patients could opt to continue to receive treatment with rociletinib following radiographic progression as outlined in the National Comprehensive Cancer Network (NCCN) guidelines for treatment of NSCLC with EGFR-TKIs if the patient provided consent, and the investigator and sponsor approved.
- Rociletinib 900 mg BID FB Capsules: Rociletinib free base (FB) dose 900 mg twice a day (BID). Rociletinib FB capsules were administered in Phase 1 only (until November 2013) and were provided in 50 mg or 150 mg white capsules. Patients were instructed to take each dose with 8 oz (240 mL) of water and with a meal or within 30 minutes after a meal. Patients received rociletinib in 21-day treatment cycles and were treated until there was progression by RECIST v1.1, clinical tumor progression, or unacceptable toxicity, or other discontinuation criteria were met. Patients could opt to continue to receive treatment with rociletinib following radiographic progression as outlined in the National Comprehensive Cancer Network (NCCN) guidelines for treatment of NSCLC with EGFR-TKIs if the patient provided consent, and the investigator and sponsor approved.
- Rociletinib 500 mg BID HBr Tablets: Rociletinib hydrobromide (HBr) dose 500 mg twice a day (BID). Rociletinib hydrobromide (HBr) tablets were administered in Phase 1 (starting in August 2013) and in all Phase 2 cohorts and were provided in 50 mg or 150 mg white capsules. Patients were instructed to take each dose with 8 oz (240 mL) of water and with a meal or within 30 minutes after a meal. Patients received rociletinib in 21-day cycles and were treated until there was progression by RECIST v1.1, clinical tumor progression, or unacceptable toxicity, or other discontinuation criteria were met. Patients could opt to continue to receive treatment with rociletinib following radiographic progression as outlined in the National Comprehensive Cancer Network (NCCN) guidelines for treatment of NSCLC with EGFR-TKIs if the patient provided consent, and the investigator and sponsor approved.
- Rociletinib 625 mg BID HBr Tablets: Rociletinib hydrobromide (HBr) dose 625 mg twice a day (BID). Rociletinib hydrobromide (HBr) tablets were administered in Phase 1 (starting in August 2013) and in all Phase 2 cohorts and were provided in 50 mg or 150 mg white capsules. Patients were instructed to take each dose with 8 oz (240 mL) of water and with a meal or within 30 minutes after a meal. Patients received rociletinib in 21-day cycles and were treated until there was progression by RECIST v1.1, clinical tumor progression, or unacceptable toxicity, or other discontinuation criteria were met. Patients could opt to continue to receive treatment with rociletinib following radiographic progression as outlined in the National Comprehensive Cancer Network (NCCN) guidelines for treatment of NSCLC with EGFR-TKIs if the patient provided consent, and the investigator and sponsor approved.
- Rociletinib 750 mg BID HBr Tablets: Rociletinib hydrobromide (HBr) dose 750 mg twice a day (BID). Rociletinib hydrobromide (HBr) tablets were administered in Phase 1 (starting in August 2013) and in all Phase 2 cohorts and were provided in 50 mg or 150 mg white capsules. Patients were instructed to take each dose with 8 oz (240 mL) of water and with a meal or within 30 minutes after a meal. Patients received rociletinib in 21-day cycles and were treated until there was progression by RECIST v1.1, clinical tumor progression, or unacceptable toxicity, or other discontinuation criteria were met. Patients could opt to continue to receive treatment with rociletinib following radiographic progression as outlined in the National Comprehensive Cancer Network (NCCN) guidelines for treatment of NSCLC with EGFR-TKIs if the patient provided consent, and the investigator and sponsor approved.
- Rociletinib 1000 mg BID HBr Tablets: Rociletinib hydrobromide (HBr) dose 1000 mg twice a day (BID). Rociletinib hydrobromide (HBr) tablets were administered in Phase 1 (starting in August 2013) and in all Phase 2 cohorts and were provided in 50 mg or 150 mg white capsules. Patients were instructed to take each dose with 8 oz (240 mL) of water and with a meal or within 30 minutes after a meal. Patients received rociletinib in 21-day cycles and were treated until there was progression by RECIST v1.1, clinical tumor progression, or unacceptable toxicity, or other discontinuation criteria were met. Patients could opt to continue to receive treatment with rociletinib following radiographic progression as outlined in the National Comprehensive Cancer Network (NCCN) guidelines for treatment of NSCLC with EGFR-TKIs if the patient provided consent, and the investigator and sponsor approved.
Period: Overall Study
Arm/Group | Rociletinib <900 mg BID FB Capsules | Rociletinib 900 mg BID FB Capsules | Rociletinib 500 mg BID HBr Tablets | Rociletinib 625 mg BID HBr Tablets | Rociletinib 750 mg BID HBr Tablets | Rociletinib 1000 mg BID HBr Tablets
Started (Total) | 38 | 19 | 209 | 245 | 95 | 6
Started Phase 1 (Upon completion of Cycle 1, Phase 1 pts could participate in an optional Treatment-extension Period) | 38 | 19 | 18 | 17 | 13 | 6
Started Phase 2 | 0 | 0 | 191 | 228 | 82 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 38 | 19 | 209 | 245 | 95 | 6
Not completed — Progressive Disease | 35 | 17 | 150 | 182 | 76 | 4
Not completed — Adverse Event | 2 | 1 | 29 | 40 | 13 | 2
Not completed — Death | 0 | 0 | 3 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 13 | 11 | 3 | 0
Not completed — Physician Decision | 0 | 0 | 2 | 5 | 0 | 0
Not completed — Other Reason | 0 | 1 | 11 | 4 | 1 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Protocol Deviation | 0 | 0 | 0 | 2 | 0 | 0
Not completed — Missing | 0 | 0 | 1 | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Rociletinib <900 mg BID FB Capsules: Rociletinib free base (FB) dose <900 mg twice a day (BID).
- Rociletinib 900 mg BID FB Capsules: Rociletinib free base (FB) dose 900 mg twice a day (BID).
- Rociletinib 500 mg BID HBr Tablets: Rociletinib hydrobromide (HBr) dose 500 mg twice a day (BID).
- Rociletinib 625 mg BID HBr Tablets: Rociletinib hydrobromide (HBr) dose 625 mg twice a day (BID).
- Rociletinib 750 mg BID HBr Tablets: Rociletinib hydrobromide (HBr) dose 750 mg twice a day (BID).
- Rociletinib 1000 mg BID HBr Tablets: Rociletinib hydrobromide (HBr) dose 1000 mg twice a day (BID).
- Total: Total of all reporting groups
Arm/Group | Rociletinib <900 mg BID FB Capsules | Rociletinib 900 mg BID FB Capsules | Rociletinib 500 mg BID HBr Tablets | Rociletinib 625 mg BID HBr Tablets | Rociletinib 750 mg BID HBr Tablets | Rociletinib 1000 mg BID HBr Tablets | Total
Number analyzed (Participants) | 38 | 19 | 209 | 245 | 95 | 6 | 612
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.1 (11.54) | 58.9 (8.37) | 63.6 (11.45) | 62.5 (11.14) | 61.5 (11.82) | 65.2 (5.53) | 62.5 (11.29)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 15 | 155 | 155 | 63 | 5 | 424
  Male | 7 | 4 | 54 | 90 | 32 | 1 | 188
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 2 | 5 | 14 | 2 | 0 | 25
  Not Hispanic or Latino | 30 | 15 | 170 | 184 | 90 | 6 | 495
  Unknown or Not Reported | 6 | 2 | 34 | 47 | 3 | 0 | 92
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 1 | 0 | 0 | 1
  Asian | 5 | 4 | 41 | 49 | 24 | 1 | 124
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 4 | 3 | 0 | 0 | 7
  Black or African American | 0 | 0 | 7 | 8 | 2 | 0 | 17
  White | 27 | 13 | 122 | 137 | 64 | 5 | 368
  More than one race | 0 | 0 | 0 | 1 | 0 | 0 | 1
  Unknown or Not Reported | 6 | 2 | 35 | 46 | 5 | 0 | 94
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 27 | 13 | 122 | 137 | 64 | 5 | 368
  Black or African American | 0 | 0 | 7 | 8 | 2 | 0 | 17
  Asian | 5 | 4 | 41 | 49 | 24 | 1 | 124
  Other | 6 | 2 | 39 | 51 | 5 | 0 | 103
Time Since Diagnosis of NSCLC (months) [Mean (Standard Deviation); unit: Months] — Population: Data not available for one participant in the 500 mg BID Hbr treatment group.
  Months
    number analyzed (Participants) | 38 | 19 | 208 | 245 | 95 | 6 | 611
    (all) | 40.4 (29.2) | 45.4 (31.94) | 36.7 (25.81) | 36.7 (31.41) | 37.6 (29.97) | 47.4 (27.03) | 37.4 (29.17)
T790M Status ( Determined by Central Lab) [Count of Participants; unit: Participants]
  Negative | 5 | 4 | 6 | 25 | 9 | 0 | 49
  Positive | 23 | 9 | 188 | 176 | 80 | 4 | 480
  Unknown | 10 | 6 | 4 | 1 | 1 | 2 | 24
  Missing | 0 | 0 | 11 | 43 | 5 | 0 | 59
History of CNS Metastases [Count of Participants; unit: Participants] | 20 | 7 | 86 | 107 | 44 | 3 | 267
Number of Previous Therapies [Mean (Standard Deviation); unit: Therapies] | 3.8 (1.65) | 3.7 (1.66) | 2.6 (1.74) | 2.8 (1.91) | 2.9 (2.11) | 3.8 (2.04) | 2.9 (1.88)
Number of Previous TKI Therapies [Mean (Standard Deviation); unit: Therapies] | 1.7 (0.77) | 2.3 (1.48) | 1.5 (0.87) | 1.6 (0.77) | 1.6 (0.86) | 1.8 (0.75) | 1.6 (0.86)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of T790M Positive Patients With Confirmed Response Per Investigator
Description: Percentage of patients with a T790M mutation (determined by central lab) with a best overall confirmed response of partial response (PR) or complete response (CR) recorded from the start of the treatment until disease progression or recurrence. Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions, defined by and assessed as: Complete Response (CR), is disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to < 10 mm. Partial Response (PR),at least a 30% decrease in the sum of the longest diameter of target lesions, taking as reference the baseline sum of longest diameter.
Time Frame: Cycle 1 Day 1 to End of Treatment, up to approximately 42 months
Population: Intent-to-treat: All randomized patients who are confirmed by central lab to be T790M positive
Measure: Count of Participants; unit: Participants
Arm/Group | Rociletinib <900 mg BID FB Capsules | Rociletinib 900 mg BID FB Capsules | Rociletinib 500 mg BID HBr Tablets | Rociletinib 625 mg BID HBr Tablets | Rociletinib 750 mg BID HBr Tablets | Rociletinib 1000 mg BID HBr Tablets
Number analyzed (Participants) | 23 | 9 | 188 | 176 | 80 | 4
Participants | 0 | 3 | 54 | 72 | 23 | 3

2. Primary Outcome: Duration of Response (DOR) in T790M Positive Patients According to RECIST Version 1.1 as Determined by Investigator Assessment
Description: Duration of Response in patients with a T790M mutation (determined by central lab) with confirmed response per investigator. The DOR for complete response (CR) and partial response (PR) was measured from the date that any of these best responses is first recorded until the first date that progressive disease (PD) is objectively documented. For patients who continue treatment post-progression, the first date of progression was used for the analysis.
Time Frame: Cycle 1 Day 1 to End of Treatment, up to approximately 36 months
Population: The DOR was measured only in T790M positive patients with a Complete Response (CR) or Partial Response (PR). There were no responders in the Rociletinib <900 mg BID treatment group so DOR is not applicable and thus not reported.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Rociletinib 900 mg BID FB Capsules | Rociletinib 500 mg BID HBr Tablets | Rociletinib 625 mg BID HBr Tablets | Rociletinib 750 mg BID HBr Tablets | Rociletinib 1000 mg BID HBr Tablets
Number analyzed (Participants) | 3 | 54 | 72 | 23 | 3
Days | 329.0 [190.0 to 713.0] | 275.0 [226.0 to 336.0] | 274.0 [169.0 to 337.0] | 217.0 [146.0 to 340.0] | 428 [NA to NA] — There are an insufficient number of participants with events.

3. Primary Outcome: Dose Limiting Toxicity (DLT) Incidence
Description: The number of Phase 1 patients who experienced dose limiting toxicities after one cycle (21 days) of study drug.
Time Frame: Cycle 1 Day 1 to Cycle 1 Day 21
Population: The dose limiting toxicity (DLT) evaluable population includes all patients who have completed Cycle 1, and who were enrolled while the dose escalation (Phase 1) part of the study was ongoing.
Measure: Count of Participants; unit: Participants
Arm/Group | Rociletinib <900 mg BID FB Capsules | Rociletinib 900 mg BID FB Capsules | Rociletinib 500 mg BID HBr Tablets | Rociletinib 625 mg BID HBr Tablets | Rociletinib 750 mg BID HBr Tablets | Rociletinib 1000 mg BID HBr Tablets
Number analyzed (Participants) | 24 | 6 | 6 | 8 | 9 | 6
Participants | 1 | 1 | 1 | 2 | 1 | 1
Statistical Analysis 1: Comparison: Rociletinib <900 mg BID FB Capsules vs Rociletinib 900 mg BID FB Capsules vs Rociletinib 500 mg BID HBr Tablets vs Rociletinib 625 mg BID HBr Tablets vs Rociletinib 750 mg BID HBr Tablets vs Rociletinib 1000 mg BID HBr Tablets; Test type: Other; Since an MTD was never reached for any of the rociletinib FB or HBr formulations/doses, a 750 mg BID HBr starting dose was selected based on early efficacy data from Phase 1, and enrollment into Phase 2 was initiated at this dosage. As the Phase 1 efficacy data matured, the recommended dose was adjusted to 625 mg BID based on antitumor activity and safety evaluations

4. Secondary Outcome: Overall Survival (OS) Determined by Investigator Assessment
Description: Overall survival was calculated as 1+ the number of days from the first dose of study drug to death due to any cause. Patients without a documented date of death were censored on the date the patient was last known to be alive.
Time Frame: Cycle 1 Day 1 to date of death, assessed up to 42 months
Population: The overall number of patients analyzed contains centrally determined T790M positive patients only. There are 2 less patients in the <900 mg BID FB group, and 1 less patient in each of the 500, 625 and 750 mg BID dose groups because they were not followed for OS.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Rociletinib <900 mg BID FB Capsules | Rociletinib 900 mg BID FB Capsules | Rociletinib 500 mg BID HBr Tablets | Rociletinib 625 mg BID HBr Tablets | Rociletinib 750 mg BID HBr Tablets | Rociletinib 1000 mg BID HBr Tablets
Number analyzed (Participants) | 21 | 9 | 187 | 175 | 79 | 4
months | 16.3 [6.3 to 17.9] | 23.7 [1.4 to NA] — There are an insufficient number of participants with events. | 18.5 [13.0 to NA] — There are an insufficient number of participants with events. | 15.0 [12.5 to 17.3] | 12.9 [9.9 to 17.7] | 7.2 [2.2 to NA] — There are an insufficient number of participants with events.

5. Secondary Outcome: Progression Free Survival (PFS) According to RECIST Version 1.1 as Determined by Investigator Review (invPFS)
Description: Progression-free survival was calculated as the number of days from the date of the first dose of study drug to the date of disease progression or death due to any cause + 1. Patients without a documented event of disease progression were censored on the date of their last adequate tumor assessment (i.e., radiologic assessment) or date of first dose of study drug if no tumor assessments have been performed. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1), as at least a 20% increase in the sum of the longest diameter of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. The appearance of one or more new lesions is also considered progression.
Time Frame: Cycle 1 Day 1 to End of Treatment, up to approximately 42 months
Population: The overall number of patients analyzed contains centrally determined T790M positive patients only. There are 2 less patients in the <900 mg BID FB group, and 1 less patient in each of the 500 and 625 mg BID dose groups because they were not followed for PFS.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Rociletinib <900 mg BID FB Capsules | Rociletinib 900 mg BID FB Capsules | Rociletinib 500 mg BID HBr Tablets | Rociletinib 625 mg BID HBr Tablets | Rociletinib 750 mg BID HBr Tablets | Rociletinib 1000 mg BID HBr Tablets
Number analyzed (Participants) | 21 | 9 | 187 | 175 | 80 | 4
months | 2.6 [1.3 to 4.0] | 10.4 [1.4 to 12.2] | 5.7 [4.2 to 6.2] | 5.2 [4.1 to 6.2] | 4.3 [2.9 to 6.1] | 7.2 [2.2 to 16.7]

6. Secondary Outcome: PK Profile of Rociletinib - Cmax
Description: Cmax = maximum concentration following administration of rociletinib
Time Frame: Cycle 1 Day 1 to Cycle 1 Day 15, or approximately 15 days
Population: PK parameters were assessed in a subset of patients treated with rociletinib. For some parameters, the number analyzed at Day 1 and Day 15 differs from the overall number analyzed based on the number of evaluable samples collected at each time point.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Rociletinib 150 mg QD FB Capsules: Rociletinib free base (FB) dose 150 mg once a day (QD).
- Rociletinib 200 mg QD FB Capsules: Rociletinib free base (FB) dose 200 mg once a day (QD).
- Rociletinib 300 mg QD FB Capsules: Rociletinib free base (FB) dose 300 mg once a day (QD).
- Rociletinib 450 mg QD FB Capsules: Rociletinib free base (FB) dose 450 mg once a day (QD).
- Rociletinib 600 mg QD FB Capsules: Rociletinib free base (FB) dose 600 mg once a day (QD).
- Rociletinib 900 mg QD FB Capsules: Rociletinib free base (FB) dose 900 mg once a day (QD).
- Rociletinib 100 mg BID FB Capsules: Rociletinib free base (FB) dose 100 mg twice a day (BID).
- Rociletinib 300 mg BID FB Capsules: Rociletinib free base (FB) dose 300 mg twice a day (BID).
- Rociletinib 600 mg BID FB Capsules: Rociletinib free base (FB) dose 600 mg twice a day (BID).
- Rociletinib 400 mg TID FB Capsules: Rociletinib free base (FB) dose 400 mg three times a day (TID).
Arm/Group | Rociletinib 150 mg QD FB Capsules | Rociletinib 200 mg QD FB Capsules | Rociletinib 300 mg QD FB Capsules | Rociletinib 450 mg QD FB Capsules | Rociletinib 600 mg QD FB Capsules | Rociletinib 900 mg QD FB Capsules | Rociletinib 100 mg BID FB Capsules | Rociletinib 300 mg BID FB Capsules | Rociletinib 600 mg BID FB Capsules | Rociletinib 900 mg BID FB Capsules | Rociletinib 400 mg TID FB Capsules | Rociletinib 500 mg BID HBr Tablets | Rociletinib 625 mg BID HBr Tablets | Rociletinib 750 mg BID HBr Tablets | Rociletinib 1000 mg BID HBr Tablets
Number analyzed (Participants) | 9 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 5 | 19 | 3 | 18 | 21 | 23 | 6
ng/mL
  Day 1 Cmax | 537 (71) | 533 (63) | 1290 (1019) | 1800 (1224) | 969 (824) | 2470 (1482) | 574 (293) | 706 (88) | 1680 (1126) | 1650 (809) | 704 (352) | 2800 (2128) | 2980 (2235) | 2570 (1850) | 4250 (2678)
  Day 15 Cmax: number analyzed (Participants) | 8 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 5 | 19 | 3 | 16 | 16 | 22 | 5
  Day 15 Cmax | 250 (188) | 503 (377) | 1760 (1056) | 942 (857) | 981 (343) | 2200 (1100) | 729 (576) | 647 (304) | 928 (95) | 1510 (997) | 1140 (274) | 2330 (1375) | 3070 (2272) | 2100 (1029) | 2510 (728)

7. Secondary Outcome: PK Profile of Rociletinib - Tmax
Description: Tmax = time to maximum concentration following administration of rociletinib
Time Frame: Cycle 1 Day 1 to Cycle 1 Day 15, or approximately 15 days
Population: as for outcome 6
Measure: Median (Full Range); unit: Hours
Arm/Group | Rociletinib 150 mg QD FB Capsules | Rociletinib 200 mg QD FB Capsules | Rociletinib 300 mg QD FB Capsules | Rociletinib 450 mg QD FB Capsules | Rociletinib 600 mg QD FB Capsules | Rociletinib 900 mg QD FB Capsules | Rociletinib 100 mg BID FB Capsules | Rociletinib 300 mg BID FB Capsules | Rociletinib 600 mg BID FB Capsules | Rociletinib 900 mg BID FB Capsules | Rociletinib 400 mg TID FB Capsules | Rociletinib 500 mg BID HBr Tablets | Rociletinib 625 mg BID HBr Tablets | Rociletinib 750 mg BID HBr Tablets | Rociletinib 1000 mg BID HBr Tablets
Number analyzed (Participants) | 9 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 5 | 19 | 3 | 18 | 21 | 23 | 6
Hours
  Day 1 Tmax | 1.5 [1 to 2.5] | 2.5 [1 to 2.5] | 2.5 [1.5 to 6] | 1.5 [1.5 to 2.5] | 2.0 [1.5 to 2.5] | 2.5 [2.5 to 4] | 2.5 [2.5 to 4] | 4.0 [4 to 8] | 4.0 [2.5 to 6] | 4.0 [1 to 8] | 2.5 [1 to 10] | 1.5 [0.5 to 10] | 2.5 [1 to 8] | 2.5 [1 to 8] | 3.25 [1 to 4]
  Day 15 Tmax: number analyzed (Participants) | 8 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 5 | 19 | 3 | 16 | 16 | 22 | 5
  Day 15 Tmax | 2.0 [1 to 4] | 1.5 [1.5 to 2.5] | 2.5 [2.5 to 4] | 1.5 [1.5 to 2.5] | 2.5 [1.5 to 6] | 4.0 [1.5 to 4] | 2.5 [1.5 to 2.5] | 1.5 [1 to 6] | 2.5 [2.5 to 4] | 4 [0 to 8] | 10 [10 to 10] | 2.5 [1 to 8] | 2.5 [1 to 6] | 2.5 [1 to 8] | 1.5 [1 to 4]

8. Secondary Outcome: PK Profile of Rociletinib - AUC 0-24
Description: AUC 0-24 = area under the curve from 0 to 24 hours
Time Frame: Cycle 1 Day 1 to Cycle 1 Day 15, or approximately 15 days
Population: PK parameters were assessed in a subset of patients treated with rociletinib. For some parameters, the number analyzed at Day 1 and Day 15 differs from the overall number analyzed based on the number of evaluable samples collected at each time point. AUC was not calculated for patients in the 400 mg TID treatment group.
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Rociletinib 150 mg QD FB Capsules | Rociletinib 200 mg QD FB Capsules | Rociletinib 300 mg QD FB Capsules | Rociletinib 450 mg QD FB Capsules | Rociletinib 600 mg QD FB Capsules | Rociletinib 900 mg QD FB Capsules | Rociletinib 100 mg BID FB Capsules | Rociletinib 300 mg BID FB Capsules | Rociletinib 600 mg BID FB Capsules | Rociletinib 900 mg BID FB Capsules | Rociletinib 500 mg BID HBr Tablets | Rociletinib 625 mg BID HBr Tablets | Rociletinib 750 mg BID HBr Tablets | Rociletinib 1000 mg BID HBr Tablets
Number analyzed (Participants) | 9 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 5 | 19 | 18 | 21 | 23 | 6
ng*hr/mL
  Day 1 AUC 0-24: number analyzed (Participants) | 9 | 2 | 3 | 3 | 3 | 3 | 3 | 3 | 5 | 18 | 16 | 20 | 19 | 6
  Day 1 AUC 0-24 | 2900 (290) | 5330 (5880) | 8370 (6612) | 8850 (6461) | 5840 (3387) | 13300 (6650) | 5740 (2927) | 8470 (1008) | 20400 (12444) | 16000 (8960) | 26800 (13668) | 33100 (26149) | 30300 (16968) | 50100 (35070)
  Day 15 AUC 0-24: number analyzed (Participants) | 8 | 2 | 3 | 3 | 3 | 3 | 3 | 3 | 5 | 17 | 15 | 15 | 20 | 6
  Day 15 AUC 0-24 | 1540 (970) | 3510 (2620) | 12100 (11616) | 4490 (3817) | 4800 (2256) | 11500 (6555) | 7100 (4189) | 6080 (4560) | 12100 (1404) | 17500 (10675) | 23700 (13035) | 31700 (18386) | 25800 (14190) | 28200 (16638)

9. Secondary Outcome: PK Profile of Rociletinib - T 1/2
Description: T 1/2 = elimination half-life following administration of rociletinib
Time Frame: Cycle 1 Day 1 to Cycle 1 Day 15, or approximately 15 days
Population: PK parameters were assessed in a subset of patients treated with rociletinib. For some parameters, the number analyzed at Day 1 and Day 15 differs from the overall number analyzed based on the number of evaluable samples collected at each time point. Elimination half-life was not calculated for patients in the 400 mg TID treatment group.
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Rociletinib 150 mg QD FB Capsules | Rociletinib 200 mg QD FB Capsules | Rociletinib 300 mg QD FB Capsules | Rociletinib 450 mg QD FB Capsules | Rociletinib 600 mg QD FB Capsules | Rociletinib 900 mg QD FB Capsules | Rociletinib 100 mg BID FB Capsules | Rociletinib 300 mg BID FB Capsules | Rociletinib 600 mg BID FB Capsules | Rociletinib 900 mg BID FB Capsules | Rociletinib 500 mg BID HBr Tablets | Rociletinib 625 mg BID HBr Tablets | Rociletinib 750 mg BID HBr Tablets | Rociletinib 1000 mg BID HBr Tablets
Number analyzed (Participants) | 9 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 5 | 19 | 18 | 21 | 23 | 6
Hours
  Day 1 T 1/2: number analyzed (Participants) | 9 | 2 | 3 | 3 | 3 | 3 | 3 | 2 | 4 | 12 | 15 | 14 | 18 | 6
  Day 1 T 1/2 | 4.8 (3.6) | 3.9 (2.3) | 4.6 (1.7) | 3.7 (1.1) | 4.4 (0.9) | 3.5 (2.8) | 3.0 (0.8) | 3.5 (1.0) | 3.6 (0.9) | 2.8 (0.7) | 2.7 (0.7) | 3.5 (1.5) | 3.1 (1.5) | 3.4 (0.9)
  Day 15 T 1/2: number analyzed (Participants) | 8 | 2 | 3 | 3 | 3 | 3 | 3 | 2 | 5 | 12 | 14 | 13 | 19 | 5
  Day 15 T 1/2 | 5.5 (3.1) | 3.5 (1.3) | 4.3 (1.2) | 3.9 (2.5) | 4.1 (2.2) | 3.5 (.56) | 3.1 (0.9) | 2.9 (0.7) | 4.7 (3.4) | 2.7 (1.9) | 3.0 (1.6) | 3.2 (0.8) | 3.6 (3.1) | 3.9 (1.9)

10. Secondary Outcome: Food Effect on PK of Rociletinib - Cmax
Description: Cmax = maximum concentration following administration of rociletinib. The effect of food on rociletinib PK parameters was assessed over a 24-hour period in blood samples from a subset of 3 patients. These patients were given a single dose of rociletinib 150mg FB 1 week prior (Day -7) to the start of continuous daily dosing after fasting. On Day 1 of Cycle 1, patients consumed a high-fat, high-calorie breakfast at the study site prior to receiving rociletinib. On each day, patients underwent blood sampling for PK at the specified time points.
Time Frame: Day -7 prior to Cycle 1 Day 1, or approximately 7 days
Population: A subset of 3 patients treated with rociletinib 150 mg FB capsules
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Cmax Fasting: Rociletinib 150 mg FB single dose given while fasting
- Cmax Fed: Rociletinib 150 mg FB single dose given with a high-fat breakfast
Arm/Group | Cmax Fasting | Cmax Fed
Number analyzed (Participants) | 3 | 3
ng/mL | 727 (354) | 1873 (2570)

11. Secondary Outcome: Food Effect on PK of Rociletinib - Tmax
Description: Tmax = time to maximum concentration following administration of rociletinib. The effect of food on rociletinib PK parameters was assessed over a 24-hour period in blood samples from a subset of 3 patients. These patients were given a single dose of rociletinib 150mg FB 1 week prior (Day -7) to the start of continuous daily dosing after fasting. On Day 1 of Cycle 1, patients consumed a high-fat, high-calorie breakfast at the study site prior to receiving rociletinib. On each day, patients underwent blood sampling for PK at the specified time points.
Time Frame: Day -7 prior to Cycle 1 Day 1, or approximately 7 days
Population: A subset of 3 patients treated with rociletinib 150 mg FB capsules
Measure: Median (Full Range); unit: Hours
Groups:
- Tmax Fasting: Rociletinib 150 mg FB single dose given while fasting
- Tmax Fed: Rociletinib 150 mg FB single dose given with a high-fat breakfast
Arm/Group | Tmax Fasting | Tmax Fed
Number analyzed (Participants) | 3 | 3
Hours | 1.5 [1.0 to 2.5] | 4.8 [2.5 to 8.0]

12. Secondary Outcome: Food Effect on PK of Rociletinib - AUC 0-24
Description: AUC 0-24 = area under the curve from 0 to 24 hours. The effect of food on rociletinib PK parameters was assessed over a 24-hour period in blood samples from a subset of 3 patients. These patients were given a single dose of rociletinib 150mg FB 1 week prior (Day -7) to the start of continuous daily dosing after fasting. On Day 1 of Cycle 1, patients consumed a high-fat, high-calorie breakfast at the study site prior to receiving rociletinib. On each day, patients underwent blood sampling for PK at the specified time points.
Time Frame: Day -7 prior to Cycle 1 Day 1, or approximately 7 days
Population: A subset of 3 patients treated with rociletinib 150 mg FB capsules. AUC could not be determined for 1 patient in the Fed arm.
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Groups:
- AUC 0-24 Fasting: Rociletinib 150 mg FB single dose given while fasting
- AUC 0-24 Fed: Rociletinib 150 mg FB single dose given with a high-fat breakfast
Arm/Group | AUC 0-24 Fasting | AUC 0-24 Fed
Number analyzed (Participants) | 3 | 2
ng*hr/mL | 4780 (3625) | 4455 (2256)

13. Secondary Outcome: Food Effect on PK of Rociletinib - C24
Description: C24 = rociletinib plasma concentration at 24 hours post the morning dose. The effect of food on rociletinib PK parameters was assessed over a 24-hour period in blood samples from a subset of 3 patients. These patients were given a single dose of rociletinib 150mg FB 1 week prior (Day -7) to the start of continuous daily dosing after fasting. On Day 1 of Cycle 1, patients consumed a high-fat, high-calorie breakfast at the study site prior to receiving rociletinib. On each day, patients underwent blood sampling for PK at the specified time points.
Time Frame: Day -7 prior to Cycle 1 Day 1, or approximately 7 days
Population: A subset of 3 patients treated with rociletinib 150 mg FB capsules
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- C24 Fasting: Rociletinib 150 mg FB single dose given while fasting
- C24 Fed: Rociletinib 150 mg FB single dose given with a high-fat breakfast
Arm/Group | C24 Fasting | C24 Fed
Number analyzed (Participants) | 3 | 3
ng/mL | 21.3 (22) | 46.5 (51)

14. Secondary Outcome: Food Effect on PK of Rociletinib - T 1/2
Description: T 1/2 = elimination half-life following administration of rociletinib. The effect of food on rociletinib PK parameters was assessed over a 24-hour period in blood samples from a subset of 3 patients. These patients were given a single dose of rociletinib 150mg FB 1 week prior (Day -7) to the start of continuous daily dosing after fasting. On Day 1 of Cycle 1, patients consumed a high-fat, high-calorie breakfast at the study site prior to receiving rociletinib. On each day, patients underwent blood sampling for PK at the specified time points.
Time Frame: Day -7 prior to Cycle 1 Day 1, or approximately 7 days
Population: A subset of 3 patients treated with rociletinib 150 mg FB capsules. Data did not allow the calculation of half-life with high fat mean in 2 patients.
Measure: Mean (Standard Deviation); unit: Hours
Groups:
- T 1/2 Fasting: Rociletinib 150 mg FB single dose given while fasting
- T 1/2 Fed: Rociletinib 150 mg FB single dose given with a high-fat breakfast
Arm/Group | T 1/2 Fasting | T 1/2 Fed
Number analyzed (Participants) | 3 | 1
Hours | 4.3 (1) | 3.1 (NA) — Data for one patient only so standard deviation not applicable.

15. Secondary Outcome: QTcF Values Post Baseline by Daily Dose
Description: Frequency of QT interval prolongation by daily dose (corrected using Fridericia's method, QTcF). To evaluate the effects of rociletinib on the QT (interval from Q wave to T wave)/QTc (interval corrected for heart rate) interval, all patients underwent serial ECG monitoring at Baseline, on Cycle 1 Day 1, Cycle 1 Day 15, on Day 1 of all subsequent cycles, at the EOT Visit, and as clinically indicated. Worst post-baseline QTcF value was used to categorize each patient.
Time Frame: Screening to End of Treatment, up to approximately 42 months
Population: Safety population by daily dose
Measure: Count of Participants; unit: Participants
Arm/Group | Rociletinib <900 mg BID FB Capsules | Rociletinib 900 mg BID FB Capsules | Rociletinib 500 mg BID HBr Tablets | Rociletinib 625 mg BID HBr Tablets | Rociletinib 750 mg BID HBr Tablets | Rociletinib 1000 mg BID HBr Tablets
Number analyzed (Participants) | 38 | 19 | 209 | 245 | 95 | 6
Participants
  QTcF Post-Baseline <450 msec | 34 | 10 | 93 | 99 | 35 | 2
  QTcF Post-Baseline 450-480 msec | 4 | 7 | 71 | 93 | 30 | 2
  QTcF Post-Baseline 481-500 msec | 0 | 1 | 23 | 24 | 11 | 2
  QTcF Post-Baseline >=501 msec | 0 | 1 | 22 | 29 | 19 | 0

16. Secondary Outcome: QTcF Value Change From Baseline
Description: QTcF value change from baseline by daily dose (corrected using Fridericia's method, QTcF). To evaluate the effects of rociletinib on the QT (interval from Q wave to T wave)/QTc (interval corrected for heart rate) interval, all patients underwent serial ECG monitoring at Baseline, on Cycle 1 Day 1, Cycle 1 Day 15, on Day 1 of all subsequent cycles, at the EOT Visit, and as clinically indicated. Worst post-baseline QTcF value was used to categorize each patient.
Time Frame: Screening to End of Treatment, up to approximately 42 months
Population: Safety population by daily dose
Measure: Count of Participants; unit: Participants
Arm/Group | Rociletinib <900 mg BID FB Capsules | Rociletinib 900 mg BID FB Capsules | Rociletinib 500 mg BID HBr Tablets | Rociletinib 625 mg BID HBr Tablets | Rociletinib 750 mg BID HBr Tablets | Rociletinib 1000 mg BID HBr Tablets
Number analyzed (Participants) | 38 | 19 | 209 | 245 | 95 | 6
Participants
  QTcF Change from Baseline <=30 msec | 29 | 11 | 47 | 55 | 12 | 1
  QTcF Change from Baseline 30-60 msec | 9 | 8 | 104 | 101 | 39 | 3
  QTcF Change from Baseline >60 msec | 0 | 0 | 58 | 89 | 44 | 2

17. Secondary Outcome: Objective Response Rate (ORR), Duration of Response (DOR) and Progression-Free Survival (PFS) Per RECIST Version 1.1 as Determined by IRR
Description: Objective response rate (ORR), duration of response (DOR) and progression-free survival (PFS) per RECIST Version 1.1 as determined by independent radiology review (IRR)
Time Frame: Cycle 1 Day 1 to End of Treatment / End of Follow-up
Population: Tumor scans were collected for independent evaluation, however ORR, DOR and PFS analyses were not performed by the central reader since the sponsor deemed not necessary following early study termination. Therefore, all IRR outcome measures were not collected and can not be reported.
Arm/Group | Rociletinib 500 mg BID HBr Tablets | Rociletinib 625 mg BID HBr Tablets
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were reported from the date of first dose of study drug and within 28 days after last dose of study drug, or up to approximately 42 months. In addition, study procedure-related AEs that occur after signing of the informed consent form and before first dose of study drug were expected to be reported. Any Serious Adverse Events or Adverse Events of Special Interest were followed until resolution or stabilization, or until patient is lost to follow-up.
Description: If a subject experiences the same preferred term (system organ class) multiple times, then the subject will be counted only once for that preferred term (system organ class).
Arm/Group | Rociletinib <900 mg BID FB Capsules | Rociletinib 900 mg BID FB Capsules | Rociletinib 500 mg BID HBr Tablets | Rociletinib 625 mg BID HBr Tablets | Rociletinib 750 mg BID HBr Tablets | Rociletinib 1000 mg BID HBr Tablets
All-Cause Mortality (participants affected / at risk) | 4/38 | 4/19 | 31/209 | 40/245 | 19/95 | 3/6
Serious Adverse Events (participants affected / at risk) | 14/38 | 8/19 | 106/209 | 138/245 | 54/95 | 5/6
Other Adverse Events (participants affected / at risk) | 37/38 | 19/19 | 208/209 | 244/245 | 95/95 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Rociletinib <900 mg BID FB Capsules (N=38) | Rociletinib 900 mg BID FB Capsules (N=19) | Rociletinib 500 mg BID HBr Tablets (N=209) | Rociletinib 625 mg BID HBr Tablets (N=245) | Rociletinib 750 mg BID HBr Tablets (N=95) | Rociletinib 1000 mg BID HBr Tablets (N=6)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 4 | 2 | 2 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1 | 1 | 2 | 0
Atrial tachycardia (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0
Atrioventricular block complete (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0
Bradycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0
Cardiac arrest (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 1 | 1 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0
Pericardial effusion (Cardiac disorders) | 0 | 0 | 1 | 3 | 1 | 0
Pericarditis (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 0 | 2 | 1 | 0 | 0
Torsade de pointes (Cardiac disorders) | 0 | 0 | 0 | 2 | 0 | 0
Ventricular tachyarrhythmia (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0 | 0
Adrenal insufficiency (Endocrine disorders) | 0 | 0 | 0 | 1 | 0 | 0
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 0 | 0 | 0 | 0 | 1 | 0
Cataract (Eye disorders) | 0 | 0 | 1 | 4 | 3 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 7 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0 | 0
Ascites (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 3 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 1 | 2 | 5 | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 2 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Ileus (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0 | 0
Intestinal dilatation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Intestinal Obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Large intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 0 | 0
Mallory-Weiss syndrome (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Melaena (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 5 | 6 | 1 | 0
Oesophagitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 5 | 4 | 1 | 1
Pancreatitis acute (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Small intestinal perforation (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Subileus (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 7 | 7 | 1 | 0
Asthenia (General disorders) | 0 | 0 | 1 | 2 | 2 | 0
Fatigue (General disorders) | 0 | 0 | 2 | 1 | 0 | 1
General physical health deterioration (General disorders) | 0 | 0 | 2 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 2 | 3 | 0 | 0
Oedema peripheral (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
Pain (General disorders) | 0 | 0 | 0 | 1 | 1 | 0
Pyrexia (General disorders) | 0 | 0 | 4 | 3 | 1 | 0
Sudden death (General disorders) | 0 | 0 | 0 | 1 | 1 | 0
Bile duct obstruction (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0
Bile duct stone (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 1 | 3 | 1 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 0 | 2 | 2 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 1 | 1 | 1 | 0
Hepatic pain (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0
Liver injury (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0
Drug hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Hypersensitivity (Immune system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Arthritis bacterial (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Bacteraemia (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 2 | 0 | 1 | 0
Clostridium difficile colitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Clostridium difficile infection (Infections and infestations) | 0 | 0 | 0 | 2 | 0 | 1
Device related infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Endocarditis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Hepatic infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Influenza (Infections and infestations) | 0 | 0 | 0 | 2 | 0 | 0
Liver abscess (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Lung infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 2 | 0 | 7 | 10 | 7 | 2
Pneumonia bacterial (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Pneumonia influenzal (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Postoperative wound infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Pyelonephritis (Infections and infestations) | 0 | 0 | 0 | 2 | 0 | 0
Sepsis (Infections and infestations) | 1 | 0 | 4 | 1 | 0 | 0
Septic shock (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Serratia bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Staphylococcal bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 3 | 3 | 1 | 0
Urosepsis (Infections and infestations) | 0 | 0 | 1 | 3 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1 | 0 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0
Hip fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0
Jaw fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Radiation necrosis (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Radiation pneumonitis (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Subcutaneous haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Subdural haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Electrocardiogram QT prolonged (Investigations) | 0 | 0 | 2 | 2 | 1 | 0
Electrocardiogram T wave inversion (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
General physical condition abnormal (Investigations) | 0 | 0 | 1 | 0 | 0 | 0
Lipase increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0
Transaminases increased (Investigations) | 0 | 1 | 1 | 1 | 0 | 1
Troponin increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 2 | 7 | 1 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 | 0 | 4 | 3 | 0 | 0
Failure to thrive (Metabolism and nutrition disorders) | 0 | 0 | 2 | 0 | 0 | 0
Fluid overload (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0
Glucose tolerance impaired (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 21 | 19 | 7 | 2
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 2 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 5 | 4 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 2 | 1 | 0 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Chondrocalcinosis pyrophosphate (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 3 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 1 | 0
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 8 | 5 | 25 | 37 | 21 | 1
Malignant pleural infusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 2 | 0 | 0
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0
Metastases to skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0
Basilar artery thrombosis (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Brain oedema (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 3 | 0 | 1 | 0
Coma (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Disturbance in attention (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 1 | 2 | 0 | 0
Haemorrhage intracranial (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 1 | 2 | 3 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Seizure (Nervous system disorders) | 0 | 0 | 1 | 1 | 3 | 0
Spinal cord oedema (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Status epilepticus (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 0 | 0 | 2 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 1 | 1 | 0 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 1 | 1 | 0 | 0
Hallucination (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0
Mental status changes (Psychiatric disorders) | 0 | 0 | 0 | 0 | 2 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 2 | 1 | 1 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 2 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 1 | 1 | 0 | 0
Renal failure (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0
Pelvic pain (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0 | 0 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 8 | 10 | 0 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 1 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 5 | 2 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 0 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 2 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 4 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 3 | 5 | 1 | 0
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 0 | 0
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 3 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0
Subgaleal haematoma (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0
Venous thrombosis (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Rociletinib <900 mg BID FB Capsules (N=38) | Rociletinib 900 mg BID FB Capsules (N=19) | Rociletinib 500 mg BID HBr Tablets (N=209) | Rociletinib 625 mg BID HBr Tablets (N=245) | Rociletinib 750 mg BID HBr Tablets (N=95) | Rociletinib 1000 mg BID HBr Tablets (N=6)
Anaemia (Blood and lymphatic system disorders) | 5 | 3 | 47 | 74 | 19 | 1
Increased tendency to bruise (Blood and lymphatic system disorders) | 0 | 2 | 1 | 0 | 1 | 0
Leukocytosis (Blood and lymphatic system disorders) | 2 | 0 | 3 | 3 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 1 | 0 | 8 | 8 | 6 | 0
Lymphopenia (Blood and lymphatic system disorders) | 0 | 1 | 9 | 9 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 10 | 11 | 7 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 3 | 3 | 21 | 19 | 17 | 0
Sinus tachycardia (Cardiac disorders) | 1 | 1 | 10 | 1 | 2 | 0
Deafness unilateral (Ear and labyrinth disorders) | 0 | 1 | 1 | 0 | 0 | 0
Dysacusis (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0 | 0
Cataract (Eye disorders) | 0 | 0 | 16 | 29 | 17 | 2
Diplopia (Eye disorders) | 0 | 1 | 2 | 1 | 0 | 0
Dry eye (Eye disorders) | 1 | 1 | 4 | 9 | 0 | 0
Lacrimation increased (Eye disorders) | 0 | 1 | 0 | 2 | 0 | 0
Vision blurred (Eye disorders) | 1 | 1 | 13 | 18 | 13 | 0
Visual acuity reduced (Eye disorders) | 1 | 1 | 4 | 2 | 0 | 0
Visual impairment (Eye disorders) | 0 | 0 | 5 | 5 | 3 | 1
Vitreous floaters (Eye disorders) | 0 | 1 | 3 | 1 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 1 | 8 | 8 | 3 | 0
Abdominal pain (Gastrointestinal disorders) | 3 | 4 | 25 | 39 | 17 | 0
Abdominal pain upper (Gastrointestinal disorders) | 2 | 0 | 15 | 18 | 11 | 2
Constipation (Gastrointestinal disorders) | 9 | 2 | 42 | 94 | 26 | 2
Diarrhoea (Gastrointestinal disorders) | 8 | 11 | 121 | 146 | 54 | 3
Dry mouth (Gastrointestinal disorders) | 2 | 0 | 26 | 22 | 16 | 0
Dyspepsia (Gastrointestinal disorders) | 2 | 2 | 7 | 6 | 5 | 1
Flatulence (Gastrointestinal disorders) | 0 | 1 | 3 | 3 | 2 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 2 | 22 | 26 | 12 | 0
Gingival bleeding (Gastrointestinal disorders) | 0 | 1 | 2 | 0 | 0 | 0
Ileus (Gastrointestinal disorders) | 0 | 2 | 1 | 1 | 0 | 0
Mouth ulceration (Gastrointestinal disorders) | 3 | 0 | 1 | 3 | 0 | 0
Nausea (Gastrointestinal disorders) | 14 | 11 | 95 | 138 | 51 | 3
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 5 | 5 | 1 | 1
Retching (Gastrointestinal disorders) | 0 | 1 | 3 | 0 | 1 | 0
Toothache (Gastrointestinal disorders) | 2 | 0 | 1 | 2 | 2 | 0
Vomiting (Gastrointestinal disorders) | 9 | 6 | 65 | 82 | 32 | 2
Asthenia (General disorders) | 6 | 1 | 28 | 34 | 17 | 1
Catheter site pain (General disorders) | 0 | 0 | 2 | 3 | 0 | 1
Chills (General disorders) | 1 | 1 | 6 | 9 | 1 | 0
Face oedema (General disorders) | 0 | 1 | 1 | 1 | 0 | 0
Fatigue (General disorders) | 9 | 8 | 109 | 124 | 47 | 3
Feeling abnormal (General disorders) | 0 | 1 | 1 | 0 | 1 | 0
Feeling cold (General disorders) | 1 | 0 | 2 | 0 | 1 | 1
Gait disturbance (General disorders) | 0 | 3 | 8 | 10 | 1 | 0
Influenza like illness (General disorders) | 1 | 1 | 5 | 1 | 1 | 0
Malaise (General disorders) | 0 | 1 | 5 | 3 | 2 | 0
Non-cardiac chest pain (General disorders) | 3 | 1 | 9 | 18 | 4 | 0
Oedema peripheral (General disorders) | 4 | 1 | 40 | 31 | 14 | 0
Pain (General disorders) | 1 | 1 | 7 | 8 | 6 | 0
Pyrexia (General disorders) | 4 | 2 | 19 | 27 | 7 | 0
Temperature intolerance (General disorders) | 0 | 1 | 2 | 1 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 2 | 1 | 6 | 6 | 5 | 0
Jaundice (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 0
Seasonal allergy (Immune system disorders) | 2 | 0 | 2 | 1 | 3 | 0
Bacterial disease carrier (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Candida infection (Infections and infestations) | 0 | 1 | 0 | 5 | 1 | 0
Clostridium difficile infection (Infections and infestations) | 0 | 0 | 0 | 4 | 0 | 1
Cystitis (Infections and infestations) | 0 | 1 | 3 | 1 | 0 | 0
Eye infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1
Folliculitis (Infections and infestations) | 0 | 0 | 2 | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 1 | 1 | 6 | 9 | 0 | 0
Pneumonia (Infections and infestations) | 2 | 1 | 12 | 15 | 11 | 2
Rhinitis (Infections and infestations) | 0 | 2 | 1 | 1 | 1 | 0
Sinusitis (Infections and infestations) | 0 | 1 | 6 | 9 | 1 | 0
Tooth infection (Infections and infestations) | 0 | 1 | 2 | 6 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 3 | 2 | 23 | 16 | 14 | 1
Urinary tract infection (Infections and infestations) | 1 | 1 | 27 | 25 | 18 | 0
Viral upper respiratory tract infection (Infections and infestations) | 0 | 1 | 1 | 1 | 2 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 3 | 14 | 14 | 4 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 2 | 9 | 8 | 4 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0
Hip fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 3 | 3 | 19 | 26 | 8 | 0
Amylase increased (Investigations) | 0 | 0 | 0 | 2 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 4 | 4 | 21 | 26 | 10 | 0
Blood alkaline phosphatase increased (Investigations) | 4 | 1 | 13 | 16 | 7 | 1
Blood bilirubin increased (Investigations) | 0 | 4 | 16 | 15 | 13 | 1
Blood creatinine increased (Investigations) | 0 | 2 | 13 | 20 | 7 | 1
Blood glucose increased (Investigations) | 1 | 1 | 4 | 9 | 7 | 2
Blood phosphorus decreased (Investigations) | 0 | 0 | 2 | 0 | 0 | 1
Blood urine present (Investigations) | 0 | 1 | 1 | 0 | 0 | 0
Electrocardiogram QT prolonged (Investigations) | 0 | 3 | 61 | 77 | 33 | 3
Electrocardiogram T wave abnormal (Investigations) | 0 | 1 | 0 | 0 | 1 | 0
Glycosylated haemoglobin increased (Investigations) | 0 | 1 | 2 | 12 | 2 | 1
Insulin C-peptide increased (Investigations) | 0 | 1 | 2 | 11 | 5 | 0
Lipase increased (Investigations) | 0 | 0 | 3 | 2 | 1 | 1
Lymphocyte count decreased (Investigations) | 0 | 0 | 12 | 8 | 2 | 0
Neutrophil count increased (Investigations) | 0 | 1 | 2 | 2 | 0 | 0
Platelet count decreased (Investigations) | 0 | 0 | 20 | 17 | 3 | 0
QRS axis abnormal (Investigations) | 0 | 1 | 0 | 0 | 0 | 0
Transaminases increased (Investigations) | 0 | 2 | 5 | 4 | 1 | 1
Weight decreased (Investigations) | 4 | 4 | 59 | 63 | 39 | 2
White blood cell count decreased (Investigations) | 1 | 0 | 19 | 20 | 2 | 0
Decreased appetite (Metabolism and nutrition disorders) | 9 | 10 | 80 | 92 | 43 | 4
Dehydration (Metabolism and nutrition disorders) | 3 | 4 | 21 | 30 | 12 | 0
Glucose tolerance impaired (Metabolism and nutrition disorders) | 0 | 1 | 6 | 9 | 11 | 0
Gout (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 4 | 10 | 113 | 147 | 56 | 3
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 1 | 7 | 6 | 2 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 2 | 2 | 18 | 22 | 3 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 1 | 6 | 11 | 2 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 2 | 0 | 2 | 8 | 6 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 | 27 | 44 | 14 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 25 | 30 | 10 | 2
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 2 | 25 | 24 | 8 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 | 3 | 23 | 31 | 13 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 6 | 3 | 26 | 43 | 15 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 4 | 4 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 5 | 4 | 3 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 1 | 3 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 4 | 6 | 57 | 71 | 27 | 2
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 9 | 12 | 5 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 3 | 2 | 12 | 21 | 13 | 1
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 2 | 0 | 2 | 1 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 8 | 1 | 20 | 22 | 10 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 5 | 4 | 23 | 16 | 10 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 | 0 | 14 | 23 | 5 | 0
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 11 | 5 | 28 | 38 | 26 | 1
Ageusia (Nervous system disorders) | 0 | 1 | 0 | 2 | 0 | 0
Amnesia (Nervous system disorders) | 1 | 1 | 4 | 2 | 1 | 0
Ataxia (Nervous system disorders) | 0 | 1 | 1 | 3 | 2 | 0
Balance disorder (Nervous system disorders) | 0 | 0 | 1 | 3 | 0 | 1
Disturbance in attention (Nervous system disorders) | 0 | 1 | 1 | 1 | 1 | 0
Dizziness (Nervous system disorders) | 4 | 4 | 25 | 41 | 14 | 1
Dysarthria (Nervous system disorders) | 0 | 2 | 0 | 0 | 2 | 0
Dysgeusia (Nervous system disorders) | 1 | 2 | 17 | 16 | 5 | 0
Headache (Nervous system disorders) | 6 | 5 | 57 | 57 | 20 | 1
Hemiparesis (Nervous system disorders) | 0 | 1 | 3 | 1 | 1 | 0
Hypoaesthesia (Nervous system disorders) | 1 | 3 | 5 | 6 | 2 | 0
Neuropathy peripheral (Nervous system disorders) | 1 | 1 | 5 | 9 | 4 | 0
Paraesthesia (Nervous system disorders) | 2 | 0 | 10 | 17 | 4 | 0
Restless legs syndrome (Nervous system disorders) | 0 | 1 | 0 | 0 | 1 | 0
Seizure (Nervous system disorders) | 0 | 0 | 1 | 6 | 5 | 0
Tension headache (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Tremor (Nervous system disorders) | 1 | 3 | 7 | 7 | 4 | 1
Vocal cord paralysis (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 2 | 19 | 20 | 8 | 1
Confusional state (Psychiatric disorders) | 0 | 0 | 8 | 13 | 3 | 0
Depression (Psychiatric disorders) | 3 | 3 | 8 | 12 | 4 | 1
Insomnia (Psychiatric disorders) | 4 | 2 | 19 | 31 | 8 | 0
Micturition urgency (Renal and urinary disorders) | 0 | 1 | 0 | 2 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 1 | 1 | 8 | 12 | 1 | 0
Renal impairment (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0
Urge incontinence (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0
Urinary tract disorder (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1
Apnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 9 | 3 | 62 | 59 | 15 | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 4 | 6 | 2 | 0
Dypnoea (Respiratory, thoracic and mediastinal disorders) | 10 | 2 | 51 | 65 | 20 | 2
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 12 | 9 | 7 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 7 | 12 | 2 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 3 | 12 | 1 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 6 | 7 | 2 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 6 | 7 | 2 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 8 | 7 | 1 | 0
Paranasal sinus hypersecretion (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 6 | 13 | 5 | 1
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 1 | 4 | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 7 | 3 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 5 | 6 | 2 | 1
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0 | 1 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 0 | 0
Throat tightness (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 4 | 3 | 2 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 2 | 0 | 13 | 9 | 11 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 3 | 14 | 18 | 5 | 1
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Pruritis (Skin and subcutaneous tissue disorders) | 1 | 1 | 5 | 12 | 4 | 0
Rash (Skin and subcutaneous tissue disorders) | 3 | 2 | 17 | 13 | 12 | 0
Rash morbilliform (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Skin erosion (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Flushing (Vascular disorders) | 2 | 0 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 5 | 0 | 16 | 11 | 7 | 0
Hypotension (Vascular disorders) | 0 | 1 | 4 | 9 | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All parties agree to submit all manuscripts or abstracts to all other parties 30 days prior to submission. This will enable all parties to protect proprietary information and to provide comments based on information that may not yet be available to other parties. The sponsor may request a delay in publication if there are important intellectual property concerns relating to publication, but does not have the right to suppress publication of the study results indefinitely.

DOCUMENTS (2):
  • Statistical Analysis Plan (2015-06-12): https://cdn.clinicaltrials.gov/large-docs/28/NCT01526928/SAP_000.pdf
  • Study Protocol (2016-08-03): https://cdn.clinicaltrials.gov/large-docs/28/NCT01526928/Prot_001.pdf